CLINICAL TRIAL: NCT05405816
Title: Determination of the Change in Gastroesophageal Reflux Disease After Laparoscopic Sleeve Gastrectomy by 24-hour Multichannel Intraluminal Impedance and pH Test
Brief Title: Determination of Change in Reflux Disease After Sleeve Gastrectomy by Intraluminal Impedance and pH-meter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Emre Teke, MD, assistant doctor, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: emreteke
Record Dates: First submitted 2022-05-30; First posted 2022-06-06 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Gastroesophageal Reflux Disease; Obesity, Morbid
Keywords: laparoscopic sleeve gastrectomy; Gastroesophageal reflux disease; Impedance-pH meter
MeSH Terms: conditions — Gastroesophageal Reflux; Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: Measurement of the change in gastroesophageal reflux disease after laparoscopic sleeve gastrectomy with 24-hour multichannel intraluminal impedance and pH-meter. It is aimed to determine the effect of surgery in a single group.
Who Masked: Participant, Care Provider
Masking Description: Due to the double-blind nature of the study, the outcome of the impedance procedure will not be known by the surgeon and the patient until the end of the study. Only the researcher will know the result of the impedance process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- after laparoscopic sleeve gastrectomy (Other): Patients who underwent laparoscopic sleeve gastrectomy surgery
  Interventions: Procedure: laparoscopic sleeve gastrectomy
- before laparoscopic sleeve gastrectomy surgery (No Intervention): obese patient preparing for laparoscopic sleeve gastrectomy surgery

INTERVENTIONS:
Procedure: laparoscopic sleeve gastrectomy — laparoscopic sleeve gastrectomy for obesity
  Arms: after laparoscopic sleeve gastrectomy

SUMMARY:
710 / 5.000 Çeviri sonuçları Laparoscopic sleeve gastrectomy (LSG) has become the most common bariatric procedure in obesity. The overall relationship between sleeve gastrectomy and gastroesophageal reflux disease is still unclear. Only acid reflux can be detected in the esophagus with a standard 24-hour pH-meter. A 24-hour pH-meter is normal in 30-50% of patients with nonerosive reflux. Impedance-pH meter, on the other hand, is a newly developed technique and determines all kinds of reflux (gas, liquid, acid and non-acid), the level of reflux and the clearance time of the esophagus. This prospective series aims to examine the relationship between LSG operation and esophago-gastric physiology using intraluminal impedance testing before and after LSG operation.

DETAILED DESCRIPTION:
Power analysis, Tien Yew Chern et al. (1) was based on the study conducted by As a result of the Power analysis using the G*Power program, when the effect size d (effect size): 0.834 and SD: 38.6 were taken for the reflux episode parameter, the minimum number of samples determined for Power: 0.90 and α: 0.05 was determined as n=18. Considering the data losses, the number of patients was planned as 38. A total of 20 patients were evaluated at the end of the study.

Patients over the age of 18 and younger than 64, with at least 5 years of morbid obesity (BMI >40 or >35 comorbidity), temporary or inadequate response weight loss despite dietetic-guided diet, who underwent laparoscopic sleeve gastrectomy in our clinic and wished to be included in the study were included in the study.

All patients' pre- and postoperative age, gender, weight, body mass index, comorbidities recorded in an excel file. Symptoms The F-scale for the frequency and intensity of pre- and post-operative esophageal symptoms (such as heartburn, regurgitation, epigastric pain, and bloating) will be routinely applied to patients 1 month before and 3 months after surgery. Preoperative esophagogastroscopy, which is routinely applied to all patients in our clinic, will continue to be routinely performed in the 1st month preoperatively . Esophagogastroscopy will be performed under sedation in all patients. In addition, preoperative upper abdomen USG will be performed on patients to reveal the etiology of reflux.

Twenty-four hour ambulatory combined pH-multichannel intraluminal impedance studies will be performed to document the presence of gastroesophageal reflux disease with a combined 24-Hour Multichannel Intraluminal Impedance and pHmeter. Abnormal total acid and non-acid exposure will be defined according to the 2004 consensus of Sifrim D. et al. (Gastroesophageal reflux monitoring: Review and consensus report on detection and definitions of acid, non-acid and gasreflux) (2). Patients' demeester score will be calculated routinely before and after surgery. In our study, investigators aimed to determine the preoperative and postoperative gastroesophageal disease findings of the patients by impedance, so the patients were not divided into different study groups. The diagnosis of GERD was made according to the Lyon consensus and the Update Porto consensus(3,4).The result of the impedance procedure applied to the patient will be evaluated when the study is completed. Due to the double-blind nature of the study, the outcome of the impedance procedure will not be known to the surgeon, researcher and patient who will perform the operation until the end of the study. Only the physician who performed the impedance procedure will know the result of the impedance procedure.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older and younger than 65 years.
* At least 5 years of morbid obesity (BMI >40 or >35 and comorbidity)
* Patients with transient or inadequate response weight loss despite dieting under the guidance of a dietitian.

Exclusion Criteria:

* Past upper gastrointestinal surgery,
* Paraesophageal (type 2), mixed (type 3), or sliding hiatal hernias of 3 cm or more,
* Patients with esophagitis and/or Barrett's metaplasia on upper GI endoscopy
* Those with peripheral vascular disease Those with a history of cerebrovascular accident
* Patients with coagulopathy
* History of chronic analgesic use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
24-hour multi-channel impedance ph-meter | 4 months
  Detection of reflux with 24-hour multi-channel impedance pH-meter

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih sultan mehmet training and research hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Chern TY, Chan DL, Maani J, Ferguson JS, Talbot ML. High-resolution impedance manometry and 24-hour multichannel intraluminal impedance with pH testing before and after sleeve gastrectomy: de novo reflux in a prospective series. Surg Obes Relat Dis. 2021 Feb;17(2):329-337. doi: 10.1016/j.soard.2020.09.030. Epub 2020 Sep 23. PMID 33153961
- [Background] Sifrim D, Castell D, Dent J, Kahrilas PJ. Gastro-oesophageal reflux monitoring: review and consensus report on detection and definitions of acid, non-acid, and gas reflux. Gut. 2004 Jul;53(7):1024-31. doi: 10.1136/gut.2003.033290. PMID 15194656
- [Background] Gyawali CP, Kahrilas PJ, Savarino E, Zerbib F, Mion F, Smout AJPM, Vaezi M, Sifrim D, Fox MR, Vela MF, Tutuian R, Tack J, Bredenoord AJ, Pandolfino J, Roman S. Modern diagnosis of GERD: the Lyon Consensus. Gut. 2018 Jul;67(7):1351-1362. doi: 10.1136/gutjnl-2017-314722. Epub 2018 Feb 3. PMID 29437910
- [Background] Roman S, Gyawali CP, Savarino E, Yadlapati R, Zerbib F, Wu J, Vela M, Tutuian R, Tatum R, Sifrim D, Keller J, Fox M, Pandolfino JE, Bredenoord AJ; GERD consensus group. Ambulatory reflux monitoring for diagnosis of gastro-esophageal reflux disease: Update of the Porto consensus and recommendations from an international consensus group. Neurogastroenterol Motil. 2017 Oct;29(10):1-15. doi: 10.1111/nmo.13067. Epub 2017 Mar 31. PMID 28370768